CLINICAL TRIAL: NCT01967225
Title: A Prospective, Randomized, Open-label, Active-controlled, Multicenter Study to Evaluate the Efficacy and Safety of BAY 1192631 in Japanese Patients With MRSA Infections (Skin and Soft Tissue Infection [SSTI] and SSTI-related Bacteremia)
Brief Title: Safety and Efficacy of BAY1192631 in Japanese Patients With Methicillin-resistant Staphylococcus Aureus (MRSA) Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16099
Record Dates: First submitted 2013-10-18; First posted 2013-10-22 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Skin Diseases, Infectious
Keywords: Methicillin Resistant Staphylococcus Aureus,; Skin and soft tissue infection,; Bacteremia,; Tedizolid
MeSH Terms: conditions — Skin Diseases, Infectious; Soft Tissue Infections; Bacteremia | interventions — tedizolid phosphate; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tedizolid Phosphate (Sivextro, BAY1192631) (Experimental): Participants received 200 mg BAY1192631 solution or tablet once daily (intravenous (I.V.) or oral (PO))
  Interventions: Drug: Tedizolid Phosphate (Sivextro, BAY1192631)
- Linezolid (Active Comparator): Participants received 600 mg Linezolid solution or tablet twice daily, every 12 ± 3 hours (intravenous (I.V.) or oral (PO))
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Tedizolid Phosphate (Sivextro, BAY1192631) — BAY1192631 solution or tablet 200 mg, once daily, Intravenous (IV) or By Mouth (PO) for 7-14 days for skin and soft tissue infections (SSTI) or 7-21 days for bacteremia.
  Arms: Tedizolid Phosphate (Sivextro, BAY1192631)
Drug: Linezolid — Linezolid solution or tablet 600 mg, twice daily, every 12 ±3 hours, Intravenous (IV) or By mouth (PO) 7-14 days for skin and soft tissue infections (SSTI) or 7-21 days for bacteremia.
  Arms: Linezolid

SUMMARY:
The aim of this study is to see the efficacy and safety of BAY1192631 in Japanese patients with methicillin-resistant staphylococcus aureus (MRSA) (skin and soft tissue infections (SSTI) and SSTI-related bacteremia).

ELIGIBILITY:
Inclusion Criteria

* Suspected or confirmed Methicillin-resistant Staphylococcus aureus (MRSA) infection
* Japanese Male and female patients aged 18 years or above
* Diagnosis of Skin and soft tissue infection with MRSA either suspected or confirmed as the major cause of infection, with/without SSTI (skin and soft tissue infection)-derived MRSA bacteremia suspected

Exclusion Criteria:

* Having received any systemic antibacterial potentially effective against MRSA for >/=24 hours within 3 days prior to the first infusion of a study drug, or having received/expected to receive the medication within 24 hours prior to the first infusion, unless antibacterial therapy for >/=72 hours proves to be ineffective on or lack appropriate potency (resistant) to MRSA.
* Moribund clinical condition such as death likely within the first 3 days of a study drug treatment
* History of significant allergy or intolerance to linezolid or BAY1192631
* Known or suspected human immunodeficiency virus (HIV) infection with a CD4+ T-cell count < 200/μL
* Chronic treatment with immunosuppressive drugs
* Active tuberculosis or non-tuberculous mycobacteriosis which need medical treatments
* Current or anticipated neutropenia with neutrophil count < 1,000/ mm^3
* Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) >/= 8 times the upper limit of reference range OR moderate to severe hepatic disease with Child Pugh score >/=10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-11-23 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (41):
- Japan (41):
  - Nagakute, Aichi-ken
  - Nagoya, Aichi-ken
  - Toyoake, Aichi-ken
  - Yoshida, Fukui
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Miyako-gun, Fukuoka
  - Sapporo, Hokkaido
  - Amagasaki, Hyōgo
  - Kobe, Hyōgo
  - Inashiki-gun, Ibaraki
  - Tsukuba, Ibaraki
  - Kamakura, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Kōshi, Kumamoto
  - Tsu, Mie-ken
  - Sendai, Miyagi
  - Nakagami-gun, Okinawa
  - Shimajiri, Okinawa
  - Hamamatsu, Shizuoka
  - Iwata, Shizuoka
  - Numazu, Shizuoka
  - Meguro-ku, Tokyo
  - Musashimurayama, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku-ku, Tokyo
  - Tachikawa, Tokyo
  - Yonago, Tottori
  - Shimonoseki, Yamaguchi
  - Kofu, Yamanashi
  - Fukuoka
  - Gifu
  - Kochi
  - Kumamoto
  - Nagasaki
  - Osaka
  - Shizuoka
  - Toyama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 46 study centers in Japan from 23 November 2013 (first subject, first visit) to 28 October 2016 (last subject, last visit).
Pre-assignment Details: Overall, 131 participants were screened. Among them, 6 participants failed screening. 125 participants were randomized to one of the 2 treatment groups.
Groups:
- Linezolid: Participants received 600 mg Linezolid solution or tablet twice daily, every 12 +- 3 hours (intravenous (I.V.) or oral (PO))
Period: Overall Study
Arm/Group | Tedizolid Phosphate (Sivextro, BAY1192631) | Linezolid
Started | 84 | 41
Participants Received Treatment | 83 | 41
Completed | 72 | 38
Not Completed | 12 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Switching to other therapy | 2 | 0
Not completed — Protocol driven decision point | 1 | 0
Not completed — Logistical difficulties | 1 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received treatment are analyzed for baseline characteristics.
Groups:
- Tedizolid Phosphate (Sivextro, BAY1192631) - SSTI: Participants who had skin and soft tissue infections (SSTI) including deep skin and soft tissue infection, chronic pyoderma, infection secondary to wound, burn and surgical wound, infected ulcer at baseline received 200 mg BAY1192631 solution or tablet once daily (intravenous (I.V.) or oral (PO))
- Linezoid - SSTI: Participants who had skin and soft tissue infections (SSTI) including deep skin and soft tissue infection, chronic pyoderma, infection secondary to wound, burn and surgical wound, infected ulcer at baseline received 600 mg Linezolid solution or tablet twice daily, every 12 ± 3 hours (intravenous (I.V.) or oral (PO))
- Tedizolid Phosphate (Sivextro, BAY1192631) - Bacteremia: Participants who had SSTI-related bacteremia at baseline received 200 mg BAY1192631 solution or tablet once daily (intravenous (I.V.) or oral (PO))
- Linezoid - Bacteremia: Participants who had SSTI-related bacteremia at baseline received 600 mg Linezolid solution or tablet twice daily, every 12 ± 3 hours (intravenous (I.V.) or oral (PO))
- Total: Total of all reporting groups
Arm/Group | Tedizolid Phosphate (Sivextro, BAY1192631) - SSTI | Linezoid - SSTI | Tedizolid Phosphate (Sivextro, BAY1192631) - Bacteremia | Linezoid - Bacteremia | Total
Number analyzed (Participants) | 79 | 39 | 4 | 2 | 124
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 31 | 20 | 3 | 0 | 54
  65 - 75 years | 31 | 9 | 1 | 2 | 43
  > 75 years | 17 | 10 | 0 | 0 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 12 | 2 | 1 | 42
  Male | 52 | 27 | 2 | 1 | 82
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.52 (4.70) | 25.72 (5.80) | 30.75 (11.19) | 22.35 (0.64) | 25.70 (5.34)
Lesion area [Count of Participants; unit: Participants] — Population: Lesion area is not collected or analyzed for bacteremia participants.
  Participants
    number analyzed (Participants) | 79 | 39 | 0 | 0 | 118
    <=75 cm^2 | 25 | 14 |  |  | 39
    >75 cm^2 | 54 | 25 |  |  | 79
Primary diagnosis [Count of Participants; unit: Participants]
  Deep SSTI | 44 | 22 | 0 | 0 | 66
  Chronic pyoderma | 3 | 2 | 0 | 0 | 5
  Infection secondary to wound, burn, surgical wound | 15 | 10 | 0 | 0 | 25
  Infection secondary to ulcer | 17 | 5 | 0 | 0 | 22
  Bacteremia | 0 | 0 | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at Test of Cure (TOC)
Description: Clinical response was evaluated by the masked investigator as clinical cure, clinical failure and indeterminate on the basis of the clinical symptoms/findings, vital sign and laboratory data from screening period to each evaluation point. Measurements for the assessment of clinical response included body temperature, pulse/heart rate, respiration rate, and white blood cell or band cell count.
Time Frame: 7-14 days after the end of treatment (EOT) for skin and soft tissue infections (SSTI) and 4-6 weeks after EOT for bacteremia
Population: This outcome measure was analyzed based on the microbiological evaluable population-methicillin-resistant Staphylococcus aureus (ME-MRSA) analysis set. The ME-MRSA consisted of clinical evaluable population at test of Cure (CE-TOC) analysis population who had an MRSA isolated as pathogen at the baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY1192631) - SSTI | Linezoid - SSTI | Tedizolid Phosphate (Sivextro, BAY1192631) - Bacteremia | Linezoid - Bacteremia
Number analyzed (Participants) | 29 | 10 | 0 | 2
Percentage of participants
  Clinical cure | 86.2 [75.7 to 99.1] | 80.0 |  | 0.0
  Clinical failure | 6.9 | 10.0 |  | 0.0
  Indeterminate | 6.9 | 10.0 |  | 100.0

2. Primary Outcome: Microbiological Response at Test of Cure (TOC)
Description: Microbiological response was assessed in accordance with the Guidance for the method of microbiological assessment by Japanese Chemotherapy Society.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY1192631) - SSTI | Linezoid - SSTI | Tedizolid Phosphate (Sivextro, BAY1192631) - Bacteremia | Linezoid - Bacteremia
Number analyzed (Participants) | 29 | 10 | 0 | 2
Percentage of participants
  Eradication | 93.1 | 90.0 |  | 100.0
  Persistence | 3.4 | 0.0 |  | 0.0
  Elimination(indeterminate) | 0.0 | 0.0 |  | 0.0
  Missing | 3.4 | 10.0 |  | 0.0

3. Secondary Outcome: Clinical Response at End of Treatment Visit (EOT)
Description: Clinical response was evaluated by the masked investigator as effective, ineffective and indeterminate on the basis of the clinical symptoms/findings, vital sign and laboratory data from screening period to each evaluation point. Measurements for the assessment of clinical response included body temperature, pulse/heart rate, respiration rate, and white blood cell or band cell count.
Time Frame: 7-14 days for skin and soft tissue infections (SSTI) or 7-21 days for bacteremia from the study drug administration
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY1192631) - SSTI | Linezoid - SSTI | Tedizolid Phosphate (Sivextro, BAY1192631) - Bacteremia | Linezoid - Bacteremia
Number analyzed (Participants) | 29 | 10 | 0 | 2
Percentage of participants
  Effective | 93.1 | 90.0 |  | 50.0
  Ineffective | 6.9 | 10.0 |  | 0.0
  Indeterminate | 0.0 | 0.0 |  | 50.0

4. Secondary Outcome: Microbiological Response at End of Treatment (EOT)
Description: as for outcome 2
Time Frame: 7-14 days for skin and soft tissue infections (SSTI) or 7-21 days for bacteremia from the study drug administration
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY1192631) - SSTI | Linezoid - SSTI | Tedizolid Phosphate (Sivextro, BAY1192631) - Bacteremia | Linezoid - Bacteremia
Number analyzed (Participants) | 29 | 10 | 0 | 2
Percentage of participants
  Eradication | 93.1 | 100.0 |  | 100.0
  Persistence | 6.9 | 0.0 |  | 0.0
  Elimination (indeterminate) | 0.0 | 0.0 |  | 0.0

5. Secondary Outcome: Change of the Lesion Size From the Screening Visit by Visit (Only Skin and Soft Tissue Infection [SSTI])
Description: Lesion size was measured by the masked investigators of erythema, edema, or induration whichever is largest.
Time Frame: Multiple time points up to 7-14 days after the end of treatment
Population: This outcome measure was analyzed based on the microbiological evaluable population-ME-MRSA analysis set. The ME-MRSA consisted of clinical evaluable population at test of Cure (CE-TOC) analysis population who had an MRSA isolated as pathogen at the baseline. Data of SSTI target participants were reported for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Tedizolid Phosphate (Sivextro, BAY1192631) - SSTI | Linezoid - SSTI
Number analyzed (Participants) | 29 | 10
cm^2
  Day 3/4 | -62.05 (96.89) | -173.93 (210.19)
  Day 5 to 13: number analyzed (Participants) | 20 | 8
  Day 5 to 13 | -134.31 (153.3) | -317.66 (410.86)
  End of treatment | -174.96 (283.05) | -280.69 (386.64)
  Test of cure (n=28, 9): number analyzed (Participants) | 28 | 9
  Test of cure (n=28, 9) | -212.63 (369.43) | -314.18 (402.93)

6. Secondary Outcome: Reduction Ratio of the Lesion Size From the Screening Visit to Day 3 to Day 4 Visit (Only Skin and Soft Tissue Infection [SSTI])
Description: Lesion size was measured by the masked investigators of erythema, edema, or induration whichever is largest. Reduction ratio (%) = 100 * (the post baseline value - baseline value) / baseline value. Negative values represent reduction of lesion size compared to baseline.
Time Frame: Baseline and Day 3/4, Day 5/13, EOT, TOC
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Tedizolid Phosphate (Sivextro, BAY1192631) - SSTI | Linezoid - SSTI
Number analyzed (Participants) | 29 | 10
Percentage
  Day3/4 | -32.32 (40.50) | -61.46 (33.31)
  Day 5 to 13: number analyzed (Participants) | 20 | 8
  Day 5 to 13 | -53.30 (41.66) | -94.61 (6.32)
  End of Treatment | -67.69 (32.40) | -90.09 (26.38)
  Test of Cure: number analyzed (Participants) | 28 | 9
  Test of Cure | -81.82 (23.99) | -99.09 (2.08)

ADVERSE EVENTS:
Time Frame: 25 days after the last study medication administration
Arm/Group | Tedizolid Phosphate (Sivextro, BAY1192631) | Linezolid
Serious Adverse Events (participants affected / at risk) | 7/83 | 4/41
Other Adverse Events (participants affected / at risk) | 64/83 | 31/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tedizolid Phosphate (Sivextro, BAY1192631) (N=83) | Linezolid (N=41)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Gas gangrene (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1)
Sternitis (Infections and infestations) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tedizolid Phosphate (Sivextro, BAY1192631) (N=83) | Linezolid (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 4 (4)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (5)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (7) | 4 (6)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (2)
Decreased activity (General disorders) | 0 (0) | 1 (1)
Injection site dermatitis (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 4 (5) | 0 (0)
Injection site hypersensitivity (General disorders) | 1 (2) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 1 (2)
Injection site pain (General disorders) | 5 (7) | 4 (4)
Injection site phlebitis (General disorders) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0)
Instillation site pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (2)
Injection site swelling (General disorders) | 3 (3) | 1 (1)
Infusion site extravasation (General disorders) | 2 (2) | 0 (0)
Puncture site pain (General disorders) | 3 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 3 (3)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (5) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Blood potassium decreased (Investigations) | 1 (2) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 1 (2)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 3 (3) | 2 (2)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Band neutrophil percentage increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 2 (2)
Liver function test increased (Investigations) | 3 (3) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (11) | 2 (4)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Asteatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 0 (0)
Vascular pain (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days